CLINICAL TRIAL: NCT01744730
Title: Safety and Pharmacokinetics of Multiple-Dose Intravenous and Oral Clindamycin in Pediatric Subjects With BMI ≥ 85th Percentile (NICHD): CLIN01
Brief Title: Safety and Pharmacokinetics of Clindamycin in Pediatric Subjects With BMI ≥ 85th Percentile
Acronym: CLIN01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Phillip Brian Smith (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor-Investigator, Phillip Brian Smith, Associate Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00041855; HHSN275201000003I (Other: National Institute of Child Health & Human Development)
Record Dates: First submitted 2012-12-05; First posted 2012-12-07 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-10

CONDITIONS: Bacterial Infections; Obesity
Keywords: Bacterial infections; Obesity; pharmacokinetics; clindamycin
MeSH Terms: conditions — Bacterial Infections; Obesity | interventions — Clindamycin; clindamycin phosphate; clindamycin palmitate; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Clindamycin IV-ages 2 to 11 Years Old (BMI 85-95th Percentile) (Active Comparator): Clindamycin IV: Children ages 2 to 11 years old with BMI 85th to 95th percentile. Their schedule of IV Clindamycin administration included 30-40 mg/kg/day dosed every 6 or every 8 hours with a maximum daily dose of 2.7 grams/day. Dosing greater than 2.7g/day was allowed for children receiving clindamycin as part of clinical care.
  Interventions: Drug: Clindamycin
- Clindamycin IV-ages 2 to 11 Years Old (BMI Greater Than 95th) (Active Comparator): Clindamycin IV: Children ages 2 to 11 years old with BMI greater than 95th percentile. Their schedule of IV Clindamycin administration included 30-40 mg/kg/day dosed every 6 or every 8 hours with a maximum daily dose of 2.7 grams/day. Dosing greater than 2.7g/day was allowed for children receiving clindamycin as part of clinical care.
  Interventions: Drug: Clindamycin
- Clinidamycin IV-ages 12 to 17 (BMI 85-95th Percentile) (Active Comparator): Clindamycin IV: Children ages 12 to 17 years old with BMI 85th to 95th percentile. Their schedule of IV Clindamycin administration included 30-40 mg/kg/day dosed every 6 or every 8 hours with a maximum daily dose of 2.7 grams/day. Dosing greater than 2.7g/day was allowed for children receiving clindamycin as part of clinical care.
  Interventions: Drug: Clindamycin
- Clindamycin IV-ages 12 to 17 (BMI Greater Than 95th) (Active Comparator): Clindamycin IV: Children ages 12 to 17 years old with BMI greater than 95th percentile. Their schedule of IV Clindamycin administration included 30-40 mg/kg/day dosed every 6 or every 8 hours with a maximum daily dose of 2.7 grams/day. Dosing greater than 2.7g/day was allowed for children receiving clindamycin as part of clinical care.
  Interventions: Drug: Clindamycin

INTERVENTIONS:
Drug: Clindamycin — Schedule includes 30-40 mg/kg/day dosed every 6 or every 8 hours with a maximum daily dose of 2.7 grams/day. Dosing greater than 2.7g/day will be allowed for children receiving clindamycin as part of clinical care.
  Other Names: Clindamycin phosphate (intravenous); Clindamycin hydrochloride (oral capsules); Clindamycin palmitate (oral solution)

SUMMARY:
The purpose of this study is to better understand how clindamycin works in children who fall in the 85th percentile or higher for body mass index (BMI - a ratio of weight to height). The results of the study will help better understand if children in higher BMI ranges process the medication differently and whether dosing should be adjusted in these children.

DETAILED DESCRIPTION:
This is a prospective, open-label pharmacokinetic and safety study of multiple doses of IV and oral clindamycin in overweight and obese children ages 2 to 17 years of age. The total study duration is expected to be approximately 24 months; each subject will participate in the study for up to 18 days (screening day; treatment days 1-14 [may be as short as 2 days] followed by an observation period of 3 days post discontinuation of clindamycin therapy or after day 17 (on day 18) of therapy in those who are treated with more than 14 days of clindamycin).

ELIGIBILITY:
Inclusion Criteria:

* 2 years - < 18 years of age at the time of first dose of study drug
* Suspected or confirmed infection OR receiving IV clindamycin per routine care
* Negative serum pregnancy test (if female and has reached menarche) within 24 hours of first dose of study drug and agreement to practice appropriate contraceptive measures, including abstinence, from the time of the initial pregnancy test through the last dose of study drug
* BMI ≥ 85th percentile for age and sex, based on Centers for Disease Control (CDC) recommendations
* Signed informed consent/Health Insurance Portability and Accountability Act (HIPAA) documents by the parent/legal guardian and assent (if applicable)

Exclusion Criteria:

* The following apply only to those who are NOT already receiving clindamycin per routine care:

  1. History of hypersensitivity or allergic reaction to clindamycin or lincomycin
  2. History of C. difficile colitis with previous administration of clindamycin
  3. Aspartate aminotransferase (AST) > 120 units/L
  4. Alanine aminotransferase (ALT) > 210 units/L
  5. Total bilirubin > 3 mg/dL
  6. Serum creatinine > 2 mg/dL
  7. Receiving a neuromuscular blocker as part of their therapy
* Previous participation in the study
* Subject is on prohibited medication or herbal product (see Appendix II)
* Subject is receiving extracorporeal life support (ECLS)
* Subject is post-cardiac bypass (within 24 hours)
* Subject on inotropes/pressors
* Any other condition or chronic illness that, in the opinion of the principal investigator, makes participation unadvised or unsafe

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2013-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: P. Brian Smith, MD, MHS, MPH, Principal Investigator — Duke Medical Center/Duke Clinical Research Institute; Kevin Watt, MD, Principal Investigator — Duke Medical Center/Duke Clinical Research Institute; Michael J Smith, MD, Principal Investigator — University of Louisville
Locations (4):
- United States (4):
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Mercy Hospital, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Akron Children's Hospital, Akron, Ohio

REFERENCES:
- [Background] Gerber JS, Coffin SE, Smathers SA, Zaoutis TE. Trends in the incidence of methicillin-resistant Staphylococcus aureus infection in children's hospitals in the United States. Clin Infect Dis. 2009 Jul 1;49(1):65-71. doi: 10.1086/599348. PMID 19463065
- [Background] Herigon JC, Hersh AL, Gerber JS, Zaoutis TE, Newland JG. Antibiotic management of Staphylococcus aureus infections in US children's hospitals, 1999-2008. Pediatrics. 2010 Jun;125(6):e1294-300. doi: 10.1542/peds.2009-2867. Epub 2010 May 17. PMID 20478934
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of obesity and trends in body mass index among US children and adolescents, 1999-2010. JAMA. 2012 Feb 1;307(5):483-90. doi: 10.1001/jama.2012.40. Epub 2012 Jan 17. PMID 22253364
- [Background] Kasten MJ. Clindamycin, metronidazole, and chloramphenicol. Mayo Clin Proc. 1999 Aug;74(8):825-33. doi: 10.4065/74.8.825. PMID 10473362
- [Background] Pai MP, Bearden DT. Antimicrobial dosing considerations in obese adult patients. Pharmacotherapy. 2007 Aug;27(8):1081-91. doi: 10.1592/phco.27.8.1081. PMID 17655508
- [Background] Bearden DT, Rodvold KA. Dosage adjustments for antibacterials in obese patients: applying clinical pharmacokinetics. Clin Pharmacokinet. 2000 May;38(5):415-26. doi: 10.2165/00003088-200038050-00003. PMID 10843460
- [Background] Falagas ME, Kompoti M. Obesity and infection. Lancet Infect Dis. 2006 Jul;6(7):438-46. doi: 10.1016/S1473-3099(06)70523-0. PMID 16790384
- [Background] Reed MD. Reversing the myths obstructing the determination of optimal age- and disease-based drug dosing in pediatrics. J Pediatr Pharmacol Ther. 2011 Jan;16(1):4-13. PMID 22477819
- [Background] Jacobs MR. How can we predict bacterial eradication? Int J Infect Dis. 2003 Mar;7 Suppl 1:S13-20. doi: 10.1016/s1201-9712(03)90066-x. PMID 12839703
- [Background] Bradley JS, Garonzik SM, Forrest A, Bhavnani SM. Pharmacokinetics, pharmacodynamics, and Monte Carlo simulation: selecting the best antimicrobial dose to treat an infection. Pediatr Infect Dis J. 2010 Nov;29(11):1043-6. doi: 10.1097/INF.0b013e3181f42a53. No abstract available. PMID 20975453
- [Background] Bell MJ, Shackelford P, Smith R, Schroeder K. Pharmacokinetics of clindamycin phosphate in the first year of life. J Pediatr. 1984 Sep;105(3):482-6. doi: 10.1016/s0022-3476(84)80033-5. PMID 6470871
- [Background] Koren G, Zarfin Y, Maresky D, Spiro TE, MacLeod SM. Pharmacokinetics of intravenous clindamycin in newborn infants. Pediatr Pharmacol (New York). 1986;5(4):287-92. PMID 3737273
- [Background] DeHaan RM, Schellenberg D. Clindamycin palmitate flavored granules. Multidose tolerance, absorption, and urinary excretion study in healthy children. J Clin Pharmacol New Drugs. 1972 Feb-Mar;12(2):74-83. doi: 10.1002/j.1552-4604.1972.tb00149.x. No abstract available. PMID 4480976
- [Background] DeHaan RM, Metzler CM, Schellenberg D, Vandenbosch WD. Pharmacokinetic studies of clindamycin phosphate. J Clin Pharmacol. 1973 May-Jun;13(5):190-209. doi: 10.1002/j.1552-4604.1973.tb00208.x. No abstract available. PMID 4488654
- [Background] del Carmen Carrasco-Portugal M, Lujan M, Flores-Murrieta FJ. Evaluation of gender in the oral pharmacokinetics of clindamycin in humans. Biopharm Drug Dispos. 2008 Oct;29(7):427-30. doi: 10.1002/bdd.624. PMID 18623043
- [Background] DeHaan RM, Metzler CM, Schellenberg D, VandenBosch WD, Masson EL. Pharmacokinetic studies of clindamycin hydrochloride in humans. Int J Clin Pharmacol. 1972 Jun;6(2):105-19. No abstract available. PMID 4638969
- [Background] Townsend RJ, Baker RP. Pharmacokinetic comparison of three clindamycin phosphate dosing schedules. Drug Intell Clin Pharm. 1987 Mar;21(3):279-81. doi: 10.1177/106002808702100310. PMID 3569028
- [Background] Wynalda MA, Hutzler JM, Koets MD, Podoll T, Wienkers LC. In vitro metabolism of clindamycin in human liver and intestinal microsomes. Drug Metab Dispos. 2003 Jul;31(7):878-87. doi: 10.1124/dmd.31.7.878. PMID 12814964
- [Background] Green B, Duffull S. Caution when lean body weight is used as a size descriptor for obese subjects. Clin Pharmacol Ther. 2002 Dec;72(6):743-4. doi: 10.1067/mcp.2002.129306. No abstract available. PMID 12496756
- [Background] Erstad BL. Which weight for weight-based dosage regimens in obese patients? Am J Health Syst Pharm. 2002 Nov 1;59(21):2105-10. doi: 10.1093/ajhp/59.21.2105. No abstract available. PMID 12434728
- [Background] Weiss M. How does obesity affect residence time dispersion and the shape of drug disposition curves? Thiopental as an example. J Pharmacokinet Pharmacodyn. 2008 Jun;35(3):325-36. doi: 10.1007/s10928-008-9090-8. Epub 2008 May 9. PMID 18465214
- [Background] Berezhkovskiy LM. On the accuracy of estimation of basic pharmacokinetic parameters by the traditional noncompartmental equations and the prediction of the steady-state volume of distribution in obese patients based upon data derived from normal subjects. J Pharm Sci. 2011 Jun;100(6):2482-97. doi: 10.1002/jps.22444. Epub 2011 Jan 19. PMID 21254063
- [Background] Morrish GA, Pai MP, Green B. The effects of obesity on drug pharmacokinetics in humans. Expert Opin Drug Metab Toxicol. 2011 Jun;7(6):697-706. doi: 10.1517/17425255.2011.570331. Epub 2011 Mar 22. PMID 21417960
- [Background] Leykin Y, Miotto L, Pellis T. Pharmacokinetic considerations in the obese. Best Pract Res Clin Anaesthesiol. 2011 Mar;25(1):27-36. doi: 10.1016/j.bpa.2010.12.002. PMID 21516911
- [Background] Weinstein AJ, Gibbs RS, Gallagher M. Placental transfer of clindamycin and gentamicin in term pregnancy. Am J Obstet Gynecol. 1976 Apr 1;124(7):688-91. doi: 10.1016/s0002-9378(16)33336-1. PMID 943947
- [Result] Gonzalez D, Melloni C, Yogev R, Poindexter BB, Mendley SR, Delmore P, Sullivan JE, Autmizguine J, Lewandowski A, Harper B, Watt KM, Lewis KC, Capparelli EV, Benjamin DK Jr, Cohen-Wolkowiez M; Best Pharmaceuticals for Children Act - Pediatric Trials Network Administrative Core Committee. Use of opportunistic clinical data and a population pharmacokinetic model to support dosing of clindamycin for premature infants to adolescents. Clin Pharmacol Ther. 2014 Oct;96(4):429-37. doi: 10.1038/clpt.2014.134. Epub 2014 Jun 20. PMID 24949994
- [Result] Gatti G, Flaherty J, Bubp J, White J, Borin M, Gambertoglio J. Comparative study of bioavailabilities and pharmacokinetics of clindamycin in healthy volunteers and patients with AIDS. Antimicrob Agents Chemother. 1993 May;37(5):1137-43. doi: 10.1128/AAC.37.5.1137. PMID 8517703
- See also: Pediatric Trials Network — https://pediatrictrials.org/
- See also: National Institute for Child Health and Human Development — http://www.nichd.nih.gov/Pages/index.aspx
- See also: Clindamycin Injection (Package Insert). Schaumberg, IL: APP Pharmaceuticals; 2008 — http://fresenius-kabi.us/component/productviewer/?view=search

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants (inpatients) were recruited in 4 hospitals in the United States. All participants were required to be receiving intravenous (IV) Clindamycin.
Pre-assignment Details: Patients between the ages (and inclusive of these ages) of 2 years to 17 years at time of first dose of study medication were screened for all other inclusion and exclusion criteria which includes must have body mass index (BMI) greater than or equal to 85th percentile for age and sex, based on Centers for Disease Control (CDC) recommendations.
Groups:
- Patients Less Than 21 Years of Age (NCT01431326): Standard of care clindamycin administration.
Period: Overall Study
Arm/Group | Clindamycin IV-ages 2 to 11 Years Old (BMI 85-95th Percentile) | Clindamycin IV-ages 2 to 11 Years Old (BMI Greater Than 95th) | Clinidamycin IV-ages 12 to 17 (BMI 85-95th Percentile) | Clindamycin IV-ages 12 to 17 (BMI Greater Than 95th) | Patients Less Than 21 Years of Age (NCT01431326)
Started | 4 | 3 | 4 | 11 | 178 (Please note this study (NCT01431326) is ongoing and data only represents a subset of this study.)
Completed | 4 | 3 | 4 | 11 | 178 (Please note this study (NCT01431326) is ongoing and data only represents a subset of this study.)
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clindamycin IV-ages 2 to 11 Years Old (BMI 85-95th Percentile) | Clindamycin IV-ages 2 to 11 Years Old (BMI Greater Than 95th) | Clinidamycin IV-ages 12 to 17 (BMI 85-95th Percentile) | Clindamycin IV-ages 12 to 17 (BMI Greater Than 95th) | Patients Less Than 21 Years of Age (NCT01431326) | Total
Number analyzed (Participants) | 4 | 3 | 4 | 11 | 178 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 3 | 4 | 11 | 178 | 200
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.4 (2.7) | 10.6 (1.4) | 14.6 (1.7) | 14.8 (1.7) | 7.2 (6.9) | 7.8 (6.8)
Gender [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 1 | 74 | 78
  Male | 2 | 3 | 3 | 10 | 104 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 52 | 54
  Not Hispanic or Latino | 3 | 2 | 3 | 10 | 124 | 142
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 1 | 1 | 28 | 30
  White | 4 | 2 | 2 | 10 | 132 | 150
  More than one race | 0 | 0 | 0 | 0 | 2 | 2
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 13 | 15
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 4 | 11 | NA — NCT01431326 did not collect region of enrollment. | NA — Total not calculated because data are not available (NA) in one or more arms.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Percentile] — There were fewer than 178 participants included in the analysis here. N=104 participants with available data in the Patients Less Than 21 Years of Age (NCT01431326) Arm. BMI was only calculated for children >=2y of age. As such, BMI was calculated for all 22 participants in this study but only 104/178 (58%) of participants in NCT01431326/POP01.
  Percentile | 90.5 (3.6) | 97.4 (1.2) | 91.7 (3.0) | 98.3 (1.3) | 83.1 (25.9) | 85.2 (24.1)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK) - Clearance (Cl) in Participants Who Received Multiple Doses of Intravenous (IV) Clindamycin.
Description: In order to understand the impact of obesity on clindamycin PK, PK data were combined to build a PK model from 3 studies that included both obese and non-obese children: 1) PTN_Clinda Obese study (clinicaltrials.gov/ct.gov identifier NCT01744730) n = 21; 2) PTN_POPS study (ct.gov identifier NCT01431326) n = 178; and 3) Staph Trio study (ct.gov identifier NCT01728363) n = 21. The data from the Staph-Trio study were only included for PK modeling and not intended to be compared in the analysis.
  PK sampling schedule for PTN_Clinda Obese was: Pre-dose 0 (within 15 minutes prior to IV clindamycin dose), 0.5 (± 5 minutes) after dose was administered, 1-1.5 hours (hrs) after dose, 3-4 hrs after, 5-6 hrs after, and pre-next dose. Samples were collected on multiple days and averaged to arrive at a single value. Comparison of empirical Bayesian Estimates (EBE) for clearance by age cohort are presented below.
  Sampling schedule details for PTN_POPS and Staph Trio were comparable.
Time Frame: After first study dose of IV Clindamycin through Day 14 (minimum of 3 samples; maximum of 6).
Population: In order to determine the impact of obesity and the best weight measure for dosing, only children ≥ 2 years of age were compared (PTN_Clinda obese study n = 21; PTN_POPS study n = 104; and Staph Trio study n = 0). The PK model suggested dosing should be based on Total Body Weight (TBW) regardless of obesity status.
Measure: Median (Full Range); unit: L/h
Groups:
- Clindamycin- Ages >2 to 6 Years Old (Non-Obese); Clindamycin- Ages >6 to 12 Years Old (Non-Obese); Clindamycin- Age >12 Years Old (Non-Obese): Non-obese patients were those with BMI <85th percentile.
- Clindamycin- Ages >2 to 6 Years Old (Obese); Clindamycin- Ages >6 to 12 Years Old (Obese); Clindamycin- Age >12 Years Old (Obese): Obese patients were those with BMI greater to or equal to the 85th percentile.
Arm/Group | Clindamycin- Ages >2 to 6 Years Old (Non-Obese) | Clindamycin- Ages >2 to 6 Years Old (Obese) | Clindamycin- Ages >6 to 12 Years Old (Non-Obese) | Clindamycin- Ages >6 to 12 Years Old (Obese) | Clindamycin- Age >12 Years Old (Non-Obese) | Clindamycin- Age >12 Years Old (Obese)
Number analyzed (Participants) | 8 | 12 | 15 | 20 | 26 | 44
L/h | 4.2 [0.9 to 9.1] | 5.7 [1.8 to 8.3] | 12.5 [3.6 to 34.4] | 10.7 [4.7 to 26.7] | 14.3 [5.6 to 37.4] | 19.2 [3.9 to 33.7]

2. Primary Outcome: Pharmacokinetics (PK) - Clearance (Cl) in Participants Who Received Multiple Doses of Intravenous (IV) Clindamycin.
Description: In order to understand the impact of obesity on clindamycin PK, PK data were combined to build a PK model from 3 studies that included both obese and non-obese children: 1) PTN_Clinda Obese study (clinicaltrials.gov/ct.gov identifier NCT01744730) n = 21; 2) PTN_POPS study (ct.gov identifier NCT01431326) n = 178; and 3) Staph Trio study (ct.gov identifier NCT01728363) n = 21. The data from the Staph-Trio study were only included for PK modeling and not intended to be compared in the analysis.
  PK sampling schedule for PTN_Clinda Obese was: Pre-dose 0 (within 15 minutes prior to IV clindamycin dose), 0.5 (± 5 minutes) after dose was administered, 1-1.5 hours (hrs) after dose, 3-4 hrs after, 5-6 hrs after, and pre-next dose. Samples were collected on multiple days and averaged to arrive at a single value. Comparison of EBE for clearance by age cohort normalized to 1 kg of body weight are presented below.
  Sampling schedule details for PTN_POPS and Staph Trio were comparable.
Time Frame: After first study dose of IV Clindamycin through Day 14 (minimum of 3 samples; maximum of 6 samples).
Population: as for outcome 1
Measure: Median (Full Range); unit: L/h/kg
Arm/Group | Clindamycin- Ages >2 to 6 Years Old (Non-Obese) | Clindamycin- Ages >2 to 6 Years Old (Obese) | Clindamycin- Ages >6 to 12 Years Old (Non-Obese) | Clindamycin- Ages >6 to 12 Years Old (Obese) | Clindamycin- Age >12 Years Old (Non-Obese) | Clindamycin- Age >12 Years Old (Obese)
Number analyzed (Participants) | 8 | 12 | 15 | 20 | 26 | 44
L/h/kg | 0.2 [0.1 to 0.8] | 0.3 [0.1 to 0.4] | 0.3 [0.1 to 0.8] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.5] | 0.2 [0 to 0.7]

3. Primary Outcome: Pharmacokinetics (PK) - Clearance (Cl) in Participants Who Received Multiple Doses of Intravenous (IV) Clindamycin.
Description: In order to understand the impact of obesity on clindamycin PK, PK data were combined to build a PK model from 3 studies that included both obese and non-obese children: 1) PTN_Clinda Obese study (clinicaltrials.gov/ct.gov identifier NCT01744730) n = 21; 2) PTN_POPS study (ct.gov identifier NCT01431326) n = 178; and 3) Staph Trio study (ct.gov identifier NCT01728363) n = 21. The data from the Staph-Trio study were only included for PK modeling and not intended to be compared in the analysis.
  PK sampling schedule for PTN_Clinda Obese was: Pre-dose 0 (within 15 minutes prior to IV clindamycin dose), 0.5 (± 5 minutes) after dose was administered, 1-1.5 hours (hrs) after dose, 3-4 hrs after, 5-6 hrs after, and pre-next dose. Samples were collected on multiple days and averaged to arrive at a single value. Comparison of EBE for clearance by age cohort normalized to 70 kg of body weight are presented below.
  Sampling schedule details for PTN_POPS and Staph Trio were comparable.
Time Frame: After first study dose of IV Clindamycin through Day 14 (minimum of 3 samples; maximum of 6 samples).
Population: as for outcome 1
Measure: Median (Full Range); unit: L/h/70 kg
Arm/Group | Clindamycin- Ages >2 to 6 Years Old (Non-Obese) | Clindamycin- Ages >2 to 6 Years Old (Obese) | Clindamycin- Ages >6 to 12 Years Old (Non-Obese) | Clindamycin- Ages >6 to 12 Years Old (Obese) | Clindamycin- Age >12 Years Old (Non-Obese) | Clindamycin- Age >12 Years Old (Obese)
Number analyzed (Participants) | 8 | 12 | 15 | 20 | 26 | 44
L/h/70 kg | 10.6 [3.6 to 35] | 14.8 [5.5 to 20.3] | 20.7 [7.1 to 48.5] | 14.7 [5.9 to 39.2] | 15.8 [4.7 to 34.7] | 14 [3.1 to 37.9]

4. Primary Outcome: PK - Volume of Distribution (V) in Participants Who Received Multiple Doses of Intravenous (IV) Clindamycin.
Description: In order to understand the impact of obesity on clindamycin PK, PK data were combined to build a PK model from 3 studies that included both obese and non-obese children: 1) PTN_Clinda Obese study (clinicaltrials.gov/ct.gov identifier NCT01744730) n = 21; 2) PTN_POPS study (ct.gov identifier NCT01431326) n = 178; and 3) Staph Trio study (ct.gov identifier NCT01728363) n = 21. The data from the Staph-Trio study were only included for PK modeling and not intended to be compared in the analysis.
  PK sampling schedule for PTN_Clinda Obese was: Pre-dose 0 (within 15 minutes prior to IV clindamycin dose), 0.5 (± 5 minutes) after dose was administered, 1-1.5 hours (hrs) after dose, 3-4 hrs after, 5-6 hrs after, and pre-next dose. Samples were collected on multiple days and averaged to arrive at a single value. Comparison of EBE for volume of distribution by age cohort are presented below.
  Sampling schedule details for PTN_POPS and Staph Trio were comparable.
Time Frame: After first study dose of IV Clindamycin through Day 14 (minimum of 3 samples; maximum of 6 samples).
Population: as for outcome 1
Measure: Median (Full Range); unit: L
Arm/Group | Clindamycin- Ages >2 to 6 Years Old (Non-Obese) | Clindamycin- Ages >2 to 6 Years Old (Obese) | Clindamycin- Ages >6 to 12 Years Old (Non-Obese) | Clindamycin- Ages >6 to 12 Years Old (Obese) | Clindamycin- Age >12 Years Old (Non-Obese) | Clindamycin- Age >12 Years Old (Obese)
Number analyzed (Participants) | 8 | 12 | 15 | 20 | 26 | 44
L | 15.3 [7.6 to 19.7] | 17.6 [8.4 to 25.2] | 29.0 [17.5 to 57.4] | 46.9 [32.9 to 85.8] | 60.1 [22.5 to 94.6] | 85.8 [28.5 to 160.0]

5. Post Hoc Outcome: Half-life
Description: In order to understand the impact of obesity on clindamycin PK, PK data were combined to build a PK model from 3 studies that included both obese and non-obese children: 1) PTN_Clinda Obese study (clinicaltrials.gov/ct.gov identifier NCT01744730) n = 21; 2) PTN_POPS study (ct.gov identifier NCT01431326) n = 178; and 3) Staph Trio study (ct.gov identifier NCT01728363) n = 21. The data from the Staph-Trio study were only included for PK modeling and not intended to be compared in the analysis.
  PK sampling schedule for PTN_Clinda Obese was: Pre-dose 0 (within 15 minutes prior to IV clindamycin dose), 0.5 (± 5 minutes) after dose was administered, 1-1.5 hours (hrs) after dose, 3-4 hrs after, 5-6 hrs after, and pre-next dose. Samples were collected on multiple days and averaged to arrive at a single value. Comparison of empirical Bayesian Estimates (EBE) for half-life by age cohort are presented below.
  Sampling schedule details for PTN_POPS and Staph Trio were comparable.
Time Frame: After participant transitioned from IV Clindamycin to oral Clindamycin through Day 14 (minimum of 3 samples; maximum of 6 samples).
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Clindamycin- Ages >2 to 6 Years Old (Non-Obese) | Clindamycin- Ages >2 to 6 Years Old (Obese) | Clindamycin- Ages >6 to 12 Years Old (Non-Obese) | Clindamycin- Ages >6 to 12 Years Old (Obese) | Clindamycin- Age >12 Years Old (Non-Obese) | Clindamycin- Age >12 Years Old (Obese)
Number analyzed (Participants) | 8 | 12 | 15 | 20 | 26 | 44
hours | 2.4 [1.1 to 5.9] | 2.2 [1.5 to 4.4] | 2.2 [0.9 to 5.8] | 3.0 [1.2 to 6.3] | 2.8 [1.2 to 7.6] | 3.6 [0.9 to 11.3]

6. Primary Outcome: PK - Volume of Distribution (V) in Participants Who Received Multiple Doses of Intravenous (IV) Clindamycin.
Description: In order to understand the impact of obesity on clindamycin PK, PK data were combined to build a PK model from 3 studies that included both obese & non-obese children: 1) PTN_Clinda Obese study (clinicaltrials.gov/ct.gov identifier NCT01744730) n = 21; 2) PTN_POPS study (ct.gov identifier NCT01431326) n = 178; and 3) Staph Trio study (ct.gov identifier NCT01728363) n = 21. The data from the Staph-Trio study were only included for PK modeling and not intended to be compared in the analysis.
  PK sampling schedule for PTN_Clinda Obese was: Pre-dose 0 (within 15 minutes prior to IV clindamycin dose), 0.5 (± 5 minutes) after dose was administered, 1-1.5 hours (hrs) after dose, 3-4 hrs after, 5-6 hrs after, and pre-next dose. Samples were collected on multiple days and averaged to arrive at a single value. Comparison of EBE for volume of distribution by age cohort normalized to 1kg of body weight are presented below.
  Sampling schedule details for PTN_POPS & Staph Trio were comparable.
Time Frame: After first study dose of IV Clindamycin through Day 14 (minimum of 3 samples; maximum of 6 samples).
Population: as for outcome 1
Measure: Median (Full Range); unit: L/kg
Arm/Group | Clindamycin- Ages >2 to 6 Years Old (Non-Obese) | Clindamycin- Ages >2 to 6 Years Old (Obese) | Clindamycin- Ages >6 to 12 Years Old (Non-Obese) | Clindamycin- Ages >6 to 12 Years Old (Obese) | Clindamycin- Age >12 Years Old (Non-Obese) | Clindamycin- Age >12 Years Old (Obese)
Number analyzed (Participants) | 8 | 12 | 15 | 20 | 26 | 44
L/kg | 0.8 [0.7 to 1.3] | 0.9 [0.7 to 1.0] | 0.9 [0.7 to 1.1] | 1.0 [0.7 to 1.3] | 0.9 [0.7 to 1.3] | 0.9 [0.6 to 1.6]

ADVERSE EVENTS:
Time Frame: Safety was assessed from the time of informed consent, up to 13 days after completion of the last study dose or early termination (approximately 30 days).
Groups:
- Clindamycin IV-ages 2 to 11 (BMI 85- <95th Percentile): Clindamycin IV: Children ages 2 to 11 years old with BMI 85th to <95th percentile. Their schedule of IV Clindamycin administration included 30-40 mg/kg/day dosed every 6 or every 8 hours with a maximum daily dose of 2.7 grams/day. Dosing greater than 2.7g/day was allowed for children receiving clindamycin as part of clinical care.
  Clindamycin PO: Schedule includes 30-40 mg/kg/day dosed every 6 or every 8 hours with a maximum daily dose of 2.7 g/day. Dosing greater than 2.7 g/day was allowed for children receiving clindamycin as part of clinical care.
- Clindamycin IV-ages 2 to 11 (BMI Greater Than or Equal 95th): Clindamycin IV: Children ages 2 to 11 years old with BMI greater than or equal 95th percentile. Their schedule of IV Clindamycin administration included 30-40 mg/kg/day dosed every 6 or every 8 hours with a maximum daily dose of 2.7 grams/day. Dosing greater than 2.7g/day was allowed for children receiving clindamycin as part of clinical care.
  Clindamycin PO: Schedule includes 30-40 mg/kg/day dosed every 6 or every 8 hours with a maximum daily dose of 2.7 g/day. Dosing greater than 2.7 g/day was allowed for children receiving clindamycin as part of clinical care.
- Clinidamycin IV-ages 12 to 17 (BMI 85- <95th Percentile): Clindamycin IV: Children ages 12 to 17 years old with BMI 85th to <95th percentile. Their schedule of IV Clindamycin administration included 30-40 mg/kg/day dosed every 6 or every 8 hours with a maximum daily dose of 2.7 grams/day. Dosing greater than 2.7g/day was allowed for children receiving clindamycin as part of clinical care.
  Clindamycin PO: Schedule includes 30-40 mg/kg/day dosed every 6 or every 8 hours with a maximum daily dose of 2.7 g/day. Dosing greater than 2.7 g/day was allowed for children receiving clindamycin as part of clinical care.
- Clindamycin IV-ages 12 to 17 (BMI Greater Than or Equal 95th): Clindamycin IV: Children ages 12 to 17 years old with BMI greater than or equal 95th percentile. Their schedule of IV Clindamycin administration included 30-40 mg/kg/day dosed every 6 or every 8 hours with a maximum daily dose of 2.7 grams/day. Dosing greater than 2.7g/day was allowed for children receiving clindamycin as part of clinical care.
  Clindamycin PO: Schedule includes 30-40 mg/kg/day dosed every 6 or every 8 hours with a maximum daily dose of 2.7 g/day. Dosing greater than 2.7 g/day was allowed for children receiving clindamycin as part of clinical care.
Arm/Group | Clindamycin IV-ages 2 to 11 (BMI 85- <95th Percentile) | Clindamycin IV-ages 2 to 11 (BMI Greater Than or Equal 95th) | Clinidamycin IV-ages 12 to 17 (BMI 85- <95th Percentile) | Clindamycin IV-ages 12 to 17 (BMI Greater Than or Equal 95th) | Patients Less Than 21 Years of Age (NCT01431326)
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3 | 0/4 | 0/11 | 0/178
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/4 | 2/11 | 0/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clindamycin IV-ages 2 to 11 (BMI 85- <95th Percentile) (N=4) | Clindamycin IV-ages 2 to 11 (BMI Greater Than or Equal 95th) (N=3) | Clinidamycin IV-ages 12 to 17 (BMI 85- <95th Percentile) (N=4) | Clindamycin IV-ages 12 to 17 (BMI Greater Than or Equal 95th) (N=11) | Patients Less Than 21 Years of Age (NCT01431326) (N=178)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clindamycin IV-ages 2 to 11 (BMI 85- <95th Percentile) (N=4) | Clindamycin IV-ages 2 to 11 (BMI Greater Than or Equal 95th) (N=3) | Clinidamycin IV-ages 12 to 17 (BMI 85- <95th Percentile) (N=4) | Clindamycin IV-ages 12 to 17 (BMI Greater Than or Equal 95th) (N=11) | Patients Less Than 21 Years of Age (NCT01431326) (N=178)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0

LIMITATIONS AND CAVEATS:
Data from 3 different studies was included to increase the robustness of the population PK model developed and leverage all available clindamycin PK data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No